CLINICAL TRIAL: NCT00003937
Title: Protocol for Patients With Newly-Diagnosed Non-Metastatic Osteosarcoma - A POG/CCG Pilot Intergroup Study
Brief Title: Combination Chemotherapy Plus Dexrazoxane in Treating Patients With Newly Diagnosed Nonmetastatic Osteosarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P9754; COG-P9754 (Other: Children's Oncology Group); POG-P9754 (Other: Pediatric Oncology Group); CCG-P9754 (Other: Children's Cancer Group); CDR0000067129 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Cardiac Toxicity; Sarcoma
Keywords: localized osteosarcoma; cardiac toxicity
MeSH Terms: conditions — Cardiotoxicity; Sarcoma | interventions — Cisplatin; Dexrazoxane; Razoxane; Doxorubicin; Etoposide; Ifosfamide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pilot 1 - Doxorubicin Intensification without Ifosfamide (Experimental): Dexrazoxane hydrochloride IV followed by doxorubicin hydrochloride IV plus cisplatin IV on days 1 and 2 of weeks 1 and 6. Methotrexate IV on day 1 of weeks 4, 5, 9, and 10. Patients undergo surgery on week 11. Adjuvant chemotherapy begins on day 1 of week 13. Group 1 (good response to neoadjuvant chemotherapy): Patients receive methotrexate IV over 4 hours every 3 weeks for 6 courses, beginning on week 13. Patients also receive dexrazoxane and doxorubicin hydrochloride every 3 weeks for 4 courses, beginning on week 14. Cisplatin is administered with the first 2 courses of dexrazoxane and doxorubicin. Group 2 (standard response to neoadjuvant chemotherapy): Patients receive methotrexate and cisplatin as in group 1 plus dexrazoxane and doxorubicin hydrochloride for 6 courses.
  Interventions: Drug: cisplatin; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: methotrexate; Procedure: conventional surgery
- Pilot 2 - Doxorubicin Intensification with Ifosfamide (Experimental): Preoperative therapy comprised of dexrazoxane hydrochloride, doxorubicin hydrochloride, and methotrexate as in pilot 1. Ifosfamide IV on days 1-5 of week 1. Patients undergo surgery on week 11, then begin adjuvant chemotherapy on week 13. Group 1: Patients receive methotrexate, dexrazoxane hydrochloride, and doxorubicin hydrochloride as in pilot 1, group 1. Ifosfamide is also administered on weeks 14 and 20. Cisplatin is administered on weeks 17, 23, and 26. Group 2: Patients receive methotrexate, dexrazoxane hydrochloride, and doxorubicin hydrochloride as in pilot 1, group 2. Ifosfamide is administered on weeks 14, 20, 26, and 31. Cisplatin is administered on weeks 17, 23, and 29
  Interventions: Drug: cisplatin; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: methotrexate; Procedure: conventional surgery
- Pilot 3 - Ifosfamide/Etoposide Intensification (Experimental): Preoperative therapy comprised of methotrexate, dexrazoxane hydrochloride, doxorubicin, ifosfamide, and cisplatin as in pilot 2. Patients undergo surgery on week 11, then begin adjuvant chemotherapy on week 13. Group 1: Patients receive methotrexate, dexrazoxane hydrochloride, doxorubicin, ifosfamide, and cisplatin as in pilot 2, group 1. Group 2: Patients receive methotrexate on weeks 13, 19, 29, 32, 35, and 36, high dose ifosfamide and etoposide IV over 4 hours on days 1-5 of weeks 14, 23, and 26, and cisplatin on weeks 20, 30, and 33. Dexrazoxane hydrochloride and doxorubicin hydrochloride are administered on weeks 17, 20, 30, and 33
  Interventions: Drug: cisplatin; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: methotrexate; Procedure: conventional surgery

INTERVENTIONS:
Drug: cisplatin
  Other Names: Cis-diamminedichloroplatinum II; CDDP; Platinol; NSC #119875
Drug: dexrazoxane hydrochloride
  Other Names: ADR-529; ZINECARD; ICRF-187; NSC #169780
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin; NSC #123127
Drug: etoposide
  Other Names: VP-16; VePesid; NSC #141540
  Arms: Pilot 3 - Ifosfamide/Etoposide Intensification
Drug: ifosfamide
  Other Names: IFX; IFOS; NSC #109724
  Arms: Pilot 2 - Doxorubicin Intensification with Ifosfamide; Pilot 3 - Ifosfamide/Etoposide Intensification
Drug: methotrexate
  Other Names: MTX; amethopterin; NSC #000740
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Chemoprotective drugs such as dexrazoxane may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase III trial to study the effectiveness of three combination chemotherapy regimens plus dexrazoxane in treating patients who have newly diagnosed nonmetastatic osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of three intensification regimens (doxorubicin vs doxorubicin plus ifosfamide vs doxorubicin plus ifosfamide and etoposide) in patients with newly diagnosed, previously untreated, nonmetastatic osteosarcoma. II. Determine the effect of postoperative dose intensification on outcome in patients with standard response to preoperative chemotherapy. III. Determine the effect of dexrazoxane cardioprotection during standard induction therapy on histologic response in these patients. IV. Evaluate biological factors that may predict outcome in these patients. V. Determine the safety of dexrazoxane administered with doxorubicin in combination with cisplatin or cisplatin and ifosfamide in these patients. VI. Determine the effect of dexrazoxane on cytotoxicity as measured by tumor necrosis at definitive surgery in these patients. VII. Assess the feasibility of administering doxorubicin with dexrazoxane cardioprotection or high dose ifosfamide with etoposide to standard risk patients who are also receiving methotrexate and cisplatin.

OUTLINE: This is a multicenter study. Patients are enrolled sequentially on 1 of 3 pilot intensification regimens. After surgery to completely remove the primary tumor, patients are assigned to 1 of 2 adjuvant chemotherapy groups based on percent necrosis at limb salvage. Pilot 1: (Closed to accrual as of 6/2/2000) Patients receive dexrazoxane IV followed immediately by doxorubicin IV over 20 minutes plus cisplatin IV over 4 hours on days 1 and 2 of weeks 1 and 6. Methotrexate IV over 4 hours is administered on day 1 of weeks 4, 5, 9, and 10. Patients undergo surgery on week 11. Adjuvant chemotherapy begins on day 1 of week 13. Group 1 (good response to neoadjuvant chemotherapy): Patients receive methotrexate IV over 4 hours every 3 weeks for 6 courses, beginning on week 13. Patients also receive dexrazoxane and doxorubicin every 3 weeks for 4 courses, beginning on week 14. Cisplatin is administered with the first 2 courses of dexrazoxane and doxorubicin. Group 2 (standard response to neoadjuvant chemotherapy): Patients receive methotrexate and cisplatin as in group 1 plus dexrazoxane and doxorubicin for 6 courses. Pilot 2: Patients receive preoperative therapy comprised of dexrazoxane, doxorubicin, and methotrexate as in pilot 1. Ifosfamide IV over 4 hours is also administered on days 1-5 of week 1. Patients undergo surgery on week 11, then begin adjuvant chemotherapy on week 13. Group 1: Patients receive methotrexate, dexrazoxane, and doxorubicin as in pilot 1, group 1. Ifosfamide is also administered on weeks 14 and 20. Cisplatin is administered on weeks 17, 23, and 26. Group 2: Patients receive methotrexate, dexrazoxane, and doxorubicin as in pilot 1, group 2. Ifosfamide is administered on weeks 14, 20, 26, and 31. Cisplatin is administered on weeks 17, 23, and 29. Pilot 3: (Open to accrual as of 6/2/2000) Patients receive preoperative therapy comprised of methotrexate, dexrazoxane, doxorubicin, ifosfamide, and cisplatin as in pilot 2. Patients undergo surgery on week 11, then begin adjuvant chemotherapy on week 13. Group 1: Patients receive methotrexate, dexrazoxane, doxorubicin, ifosfamide, and cisplatin as in pilot 2, group 1. Group 2: Patients receive methotrexate on weeks 13, 19, 29, 32, 35, and 36, high dose ifosfamide and etoposide IV over 4 hours on days 1-5 of weeks 14, 23, and 26, and cisplatin on weeks 20, 30, and 33. Dexrazoxane and doxorubicin are administered on weeks 17, 20, 30, and 33. Patients are followed every 3 months for 1 year, every 6 months for 4 years and then annually thereafter.

PROJECTED ACCRUAL: Approximately 180 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven newly diagnosed moderate or high grade osteosarcoma without metastases No prior treatment, including complete resection No parosteal or periosteal sarcoma No osteosarcoma associated with Paget's disease No nonresectable tumors or tumors that may result in marginal or interlesion resection Must be enrolled on protocol POG-9851

PATIENT CHARACTERISTICS: Age: 30 and under Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT no greater than 3 times normal Renal: Creatinine normal Phosphate at least 3.0 mg/dL without supplementation Cardiovascular: Shortening fraction at least 28% by echocardiogram If echocardiogram unsatisfactory, must have ejection fraction at least 50% No history of pericarditis or myocarditis No symptomatic arrhythmia or symptomatic cardiac conduction disturbances

PRIOR CONCURRENT THERAPY: See Disease Characteristics Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 253 (Actual)
Dates: Start 1999-09; Primary Completion 2004-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Schwartz, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (148):
- United States (132):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Children's Hospital and Health Center, San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Portland, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. John's Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Doernbecher Children's Hospital, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - James H. Quillen College of Medicine, Johnson City, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology P.A., Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - MBCCOP - South Texas Pediatric, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Roanoke Community Hospital, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Medical School-Charleston, Charleston, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- San Jorge Childrens Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Clinique de Pediatrie, Geneva

REFERENCES:
- [Background] Isakoff MS, Barkauskas DA, Ebb D, Morris C, Letson GD. Poor survival for osteosarcoma of the pelvis: a report from the Children's Oncology Group. Clin Orthop Relat Res. 2012 Jul;470(7):2007-13. doi: 10.1007/s11999-012-2284-9. Epub 2012 Feb 22. PMID 22354612
- [Background] Janeway KA, Barkauskas DA, Krailo MD, Meyers PA, Schwartz CL, Ebb DH, Seibel NL, Grier HE, Gorlick R, Marina N. Outcome for adolescent and young adult patients with osteosarcoma: a report from the Children's Oncology Group. Cancer. 2012 Sep 15;118(18):4597-605. doi: 10.1002/cncr.27414. Epub 2012 Jan 17. PMID 22252521
- [Derived] Kopp LM, Womer RB, Schwartz CL, Ebb DH, Franco VI, Hall D, Barkauskas DA, Krailo MD, Grier HE, Meyers PA, Wexler LH, Marina NM, Janeway KA, Gorlick R, Bernstein ML, Lipshultz SE; Children's Oncology Group. Effects of dexrazoxane on doxorubicin-related cardiotoxicity and second malignant neoplasms in children with osteosarcoma: a report from the Children's Oncology Group. Cardiooncology. 2019 Oct 28;5:15. doi: 10.1186/s40959-019-0050-9. eCollection 2019. PMID 32154021